CLINICAL TRIAL: NCT00094718
Title: Phase 1 Study of the Safety and Immunogenicity of West Nile/Dengue-4 3'delta30 Chimeric Virus Vaccine (WN/DEN4-3'delta30), a Live Attenuated Vaccine for West Nile Encephalitis
Brief Title: Safety of and Immune Response to a West Nile Virus Vaccine (WN/DEN4-3'delta30) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 206; H.22.04.10.06.A1
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: West Nile Fever Encephalitis
Keywords: Chimeric Virus Vaccine; West Nile Virus; Dengue Virus
MeSH Terms: conditions — West Nile Fever

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): One subcutaneous vaccination with WN/DEN4-3'delta30 vaccine (10^3 PFU dose) into the deltoid region of either arm.
  Interventions: Biological: WN/DEN4-3'delta30
- 2 (Experimental): One subcutaneous vaccination with WN/DEN4-3'delta30 vaccine (10^4 PFU dose) into the deltoid region of either arm. This arm may enroll after the results from Arm 1 are analyzed.
  Interventions: Biological: WN/DEN4-3'delta30
- 3 (Experimental): One subcutaneous vaccination with WN/DEN4-3'delta30 vaccine (10^5 PFU dose) into the deltoid region of either arm. This arm may enroll after the results from Arm 2 are analyzed.
  Interventions: Biological: WN/DEN4-3'delta30
- 4 (Placebo Comparator): One subcutaneous vaccination with placebo vaccine into the deltoid region of either arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: WN/DEN4-3'delta30 — Live attenuated WN/DEN4-3'delta30 vaccine (one of three doses)
  Arms: 1; 2; 3
Biological: Placebo — Placebo for WN/DEN4-3'delta30 vaccine
  Arms: 4

SUMMARY:
West Nile (WN) virus infection is an emerging disease; WN infection may lead to paralysis, coma, and death. The purpose of this study is to test the safety of and immune response to a WN vaccine in healthy adults. The vaccine is based on a live attenuated vaccine developed against dengue virus.

DETAILED DESCRIPTION:
WN is widely distributed in Africa and Europe, where it is usually associated with mild illness. In the United States, WN is considered a public health threat because severe illness caused by WN infection has caused paralysis, coma, and death, especially in the elderly. This study will evaluate the safety and immunogenicity of a live attenuated chimeric virus, WN/DEN4-3'delta30, which is derived from the DEN4 dengue virus and wild-type WN serotypes.

This study will last 180 days. Participants in Cohort 1 will be randomly assigned to receive the lowest dose of WN/DEN4-3'delta30 or placebo at study entry. Cohort 2 will begin only after safety review of all participants in Cohort 1. Participants in Cohort 2 will receive a higher dose of WN/DEN4-3'delta30 or placebo. Cohort 3 will begin only after safety review of all participants in Cohort 2. Participants in Cohort 3 will receive the highest dose of WN/DEN4-3'delta30 or placebo. Immediately after receiving their injections, participants will be observed for 30 minutes for immediate adverse reactions.

After vaccination, participants will be asked to monitor their temperatures every day for 16 days and on Day 19. Study visits will occur every other day after vaccination until Day 16, followed by 5 additional visits at selected days through Day 180. Blood collection and a targeted physical exam will occur at each study visit. Some participants will be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be followed for the duration of the study
* Willing to use acceptable methods of contraception
* Good general health

Exclusion Criteria:

* Clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Hematologic disease
* History of migraine headaches
* History of encephalitis
* Alcohol or drug abuse within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Emergency room visit or hospitalization for severe asthma within 6 months prior to study entry
* HIV-1 infected
* Hepatitis C virus infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days of study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Blood products within 6 months prior to study entry
* Participation in another investigational vaccine or drug trial within 60 days of starting this study, or while participating in this study
* Previously received a licensed or experimental yellow fever, tick-borne encephalitis, or dengue vaccine
* Surgical removal of spleen
* History of West Nile encephalitis
* History of dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus)
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2005-02; Primary Completion 2005-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Frequency of vaccine-related adverse effects, graded by severity, for each dose | Throughout study
Immunogenicity of vaccine against WN virus | Throughout study

SECONDARY OUTCOMES:
To assess the durability of the antibody response | At Day 180
To assess the frequency, quantity, and duration of viremia in each dose cohort studied | Throughout study
To assess the immunogenicity of the WN/DEN4-3'delta30 vaccine against WN wild-type virus | Throughout study
To compare the T cell medicated immune response against West Nile virus of those volunteers infected with the WN/DEN4-3'delta30 vaccine virus with that of uninfected volunteers and placebo recipients | At study completion
To evaluate the immunopathological mechanism of vaccine-associated rash in those volunteers who are willing to undergo skin biopsy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health
Locations (2):
- United States (2):
  - Johns Hopkins School of Public Health, Baltimore, Maryland
  - Vanderbilt University School of Medicine, Nashville, Tennessee

REFERENCES:
- [Background] Chang GJ, Kuno G, Purdy DE, Davis BS. Recent advancement in flavivirus vaccine development. Expert Rev Vaccines. 2004 Apr;3(2):199-220. doi: 10.1586/14760584.3.2.199. PMID 15056045
- [Background] Lai CJ, Monath TP. Chimeric flaviviruses: novel vaccines against dengue fever, tick-borne encephalitis, and Japanese encephalitis. Adv Virus Res. 2003;61:469-509. doi: 10.1016/s0065-3527(03)61013-4. PMID 14714441
- [Background] Monath TP, McCarthy K, Bedford P, Johnson CT, Nichols R, Yoksan S, Marchesani R, Knauber M, Wells KH, Arroyo J, Guirakhoo F. Clinical proof of principle for ChimeriVax: recombinant live, attenuated vaccines against flavivirus infections. Vaccine. 2002 Jan 15;20(7-8):1004-18. doi: 10.1016/s0264-410x(01)00457-1. PMID 11803060
- [Background] Pletnev AG, Claire MS, Elkins R, Speicher J, Murphy BR, Chanock RM. Molecularly engineered live-attenuated chimeric West Nile/dengue virus vaccines protect rhesus monkeys from West Nile virus. Virology. 2003 Sep 15;314(1):190-5. doi: 10.1016/s0042-6822(03)00450-1. PMID 14517072
- [Background] Pugachev KV, Guirakhoo F, Trent DW, Monath TP. Traditional and novel approaches to flavivirus vaccines. Int J Parasitol. 2003 May;33(5-6):567-82. doi: 10.1016/s0020-7519(03)00063-8. PMID 12782056